CLINICAL TRIAL: NCT04476277
Title: Red Cell Half Life Determination in Patients With and Without Sickle Cell Disease
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 200080; 20-H-0080
Record Dates: First submitted 2020-07-17; First posted 2020-07-20 (Actual); Results first posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2023-02

CONDITIONS: Sickle Cell Disease; Sickle Cell Anemia
Keywords: Red Cell Survival; Biotin; Sickle Cell Anemia; Sickle Cell Disease; Sickle Cell Trait
MeSH Terms: conditions — Anemia, Sickle Cell; Sickle Cell Trait

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Sickle Cell Disease Pre-Transplantation (Experimental): Autologous cells will be collected in participants with Sickle Cell Disease Pre-Transplantation and biotin-labeled ex vivo and reinfused to measure red cell survival
  Interventions: Drug: Biotin label
- Sickle Cell Disease Post-Transplantation (Experimental): Autologous cells will be collected in participants with Sickle Cell Disease Post-Transplantation and biotin-labeled ex vivo and reinfused to measure red cell survival
  Interventions: Drug: Biotin label
- Sickle Cell Trait (HbAS) (Experimental): Autologous cells will be collected in participants with Sickle Cell Trait (HbAS) and biotin-labeled ex vivo and reinfused to measure red cell survival
  Interventions: Drug: Biotin label
- HbAA (Healthy volunteers) (Experimental): Autologous cells will be collected in participants with HbAA (Healthy volunteers) and biotin-labeled ex vivo and reinfused to measure red cell survival
  Interventions: Drug: Biotin label

INTERVENTIONS:
Drug: Biotin label — Autologous cells will be collected and biotin-labeled ex vivo and reinfused to measure red cell survival

SUMMARY:
Background:

Sickle cell disease (SCD) is an inherited blood disorder. It results from a single genetic change (mutation) in red blood cells (RBCs). RBCs are the cells that carry oxygen to the body. In people with SCD, some RBCs are abnormal and die early. This leaves a shortage of healthy RBCs. Researchers want to learn more about how long RBCs live in the human body.

Objective:

To study how long RBCs live in people with and without SCD.

Eligibility:

People age 18 and older who either have SCD, had SCD but were cured with a bone marrow transplant, have the sickle cell trait (SCT), or are a healthy volunteer without SCD or SCT

Design:

Participants will be screened with a medical history and physical exam. They will give a blood sample.

Participants will have a small amount of blood drawn from a vein. In the laboratory, the blood will be mixed with a vitamin called biotin. Biotin sticks to the outside of RBCs without changing their function, shape, or overall lifetime. This process is known as biotin labeling of RBCs. The biotin labeled RBCs will be returned to the participant via vein injection.

Participants will give frequent blood samples. Their RBCs will be studied to see how many biotin labeled RBCs remain over time. This shows how long the RBCs live. Participants will give blood samples until no biotin labeled RBCs can be detected.

During the study visits, participants will report any major changes to their health.

Participation lasts for up to 6 months.

DETAILED DESCRIPTION:
Study Description:

This study will use biotin-labeling of red blood cells (RBCs) to determine the mean potential lifespan (MPL) of RBCs in patients with sickle cell disease (SCD) compared to patients who have successfully undergone curative bone marrow transplantation (BMT, allogeneic or autologous), participants with sickle cell trait, and healthy donors without SCD. Previous studies have corroborated the MPL of healthy donor RBCs to be approximately 115 days while RBCs from patients with SCD have a much more variable but consistently shorter MPL of approximately 32 days. Allogeneic BMT is a curative therapy for the treatment of severe SCD with stable, mixed donor recipient chimerism after BMT sufficient to reverse the sickle cell phenotype by virtue of improved donor red cell survival compared to the ineffective erythropoiesis of SCD. We predict that the hematologic variables associated with red cell survival among patients with SCD vs. participants with SCT and healthy donors can be used to determine the necessary amount of corrected hemoglobin required to overcome the red cell pathology of SCD. Data generated will be used to determine the utility of performing a population study of RBC lifespan in gene therapy treated patients to ultimately target the percentage of transferred globin gene needed to reverse SCD. The data generated will refine our understanding of the degree of correction necessary to reverse the phenotype of SCD.

Objectives:

Primary Objective: To determine and compare red blood cell survival in patients with SCD, patients with SCD who have undergone BMT, participants with SCT, and healthy donors, and validate the association of red cell survival with known markers of increased red cell survival.

Secondary Objectives: To evaluate correlation of markers of hemolysis (reticulocyte count), number of alpha globin genes, and fetal hemoglobin with RBC survival.

Endpoints:

Primary Endpoint: Red blood cell survival

Secondary Endpoints: Relationship of red blood cell survival to hematologic parameters. Antibody detection to biotin.

ELIGIBILITY:
INCLUSION CRITERIA:

* Age 18 or greater with a confirmed diagnosis of homozygous SCD (HbSS, HbSC, HbSB0), sickle cell trait (HbAS), or healthy volunteer (HbA)
* Normal renal function: creatinine <1.5 mg/dL
* Negative direct antiglobulin test (DAT)
* Ability to give informed consent to participate in the protocol

EXCLUSION CRITERIA:

* Any uncontrolled chronic illness other than sickle cell disease
* Active viral, bacterial, fungal, or parasitic infection
* Consumption of biotin supplements or raw eggs within 30 days
* Blood loss within the previous 8 weeks >540mL
* Pregnancy
* Pre-existing, naturally occurring antibodies against biotin

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2023-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John F Tisdale, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Leonard AK, Furstenau D, Inam Z, Luckett C, Chu R, Demirci S, Essawi K, Gudmundsdottir B, Hinds M, DiNicola J, Li Q, Eaton WA, Cellmer T, Wang X, Thein SL, Macari ER, VanNest S, Hsieh MM, Bonner M, Pierciey FJ, Tisdale JF. In vivo measurement of RBC survival in patients with sickle cell disease before or after hematopoietic stem cell transplantation. Blood Adv. 2024 Apr 9;8(7):1806-1816. doi: 10.1182/bloodadvances.2023011397. PMID 38181784
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2020-H-0080.html

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation | Sickle Cell Trait (HbAS) | HbAA (Healthy Volunteers)
Started | 6 | 6 | 7 | 3
Completed | 6 | 6 | 6 | 3
Not Completed | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation | Sickle Cell Trait (HbAS) | HbAA (Healthy Volunteers) | Total
Number analyzed (Participants) | 6 | 6 | 7 | 3 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 7 | 3 | 22
  >=65 years | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6 | 2 | 14
  Male | 2 | 4 | 1 | 1 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 6 | 7 | 3 | 22
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 6 | 7 | 3 | 22
  White | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 7 | 3 | 22

OUTCOME MEASURES:

1. Primary Outcome: Mean Red Blood Cells Lifespan in Participants
Description: Mean Days of Red Blood Cells (RBC) survival in participants with Sickle Cell Disease (SCD), participants with SCD who have undergone stem cell transplant, participants with Sickle Cell Trait, and healthy volunteers.
  Peripheral blood samples were analyzed by flow cytometry until biotin was not detectable on RBC.
Time Frame: Sickle Cell Disease Pre-Transplantation cohort time frame is as follows: baseline, twice weekly up to week 3 then weekly up to week 22. All other cohorts, time frame is as follows: baseline, weekly up to week 4, then every other week up to week 22.
Population: Analysis includes participants that have completed study and had no exchange or simple red blood cell transfusions.
Measure: Mean (Full Range); unit: day
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation | Sickle Cell Trait (HbAS) | HbAA (Healthy Volunteers)
Number analyzed (Participants) | 6 | 5 | 6 | 3
day | 64.1 [35 to 91] | 113.4 [105 to 119] | 126.0 [119 to 147] | 123.7 [91 to 147]
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation vs Sickle Cell Trait (HbAS) vs HbAA (Healthy Volunteers); Test type: Other; p < 0.001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Number of Participants With Antibody Detection
Description: Number of participants with Antibody detection to biotin
Time Frame: Baseline, 3 months, 6 months
Population: Analysis includes participants that have completed study and had no exchange or simple red blood cell transfusions.
Measure: Count of Participants; unit: Participants
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation | Sickle Cell Trait (HbAS) | HbAA (Healthy Volunteers)
Number analyzed (Participants) | 6 | 5 | 6 | 3
Participants | 0 | 0 | 0 | 0

3. Secondary Outcome: Mean White Blood Cell Count
Description: Mean White Blood Cell (WBC) count between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: K/mcL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
K/mcL | 9.0 (4.5) | 6.5 (2.4)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.28, t-test, 2 sided

4. Secondary Outcome: Mean Red Blood Cell Count
Description: Mean Red Blood Cell (RBC) Count between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: M/mcL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
M/mcL | 3.0 (1.0) | 4.3 (0.8)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.04, t-test, 2 sided

5. Secondary Outcome: Mean Hemoglobin Value
Description: Mean Hemoglobin (Hb) Value between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
g/dL | 8.8 (2.1) | 13.0 (2.2)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.01, t-test, 2 sided

6. Secondary Outcome: Mean Hematocrit Value
Description: Mean Hematocrit (Hct) value between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: % of Hematocrit
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
% of Hematocrit | 25.0 (6.3) | 38.3 (5.8)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.01, t-test, 2 sided

7. Secondary Outcome: Mean Value of Mean Corpuscular Volume
Description: Mean Value of Mean Corpuscular Volume (MCV) between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: fL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
fL | 86.7 (12.8) | 89.4 (2.3)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.65, t-test, 2 sided

8. Secondary Outcome: Mean Absolute Reticulocyte Count
Description: Mean Absolute Reticulocyte Count (ARC) between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: K/mcL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
K/mcL | 192.7 (84.8) | 152.9 (96.4)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.48, t-test, 2 sided

9. Secondary Outcome: Mean Aspartate Aminotransferase Value
Description: Mean Aspartate Aminotransferase (AST) value between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: IU/L
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
IU/L | 26.1 (12.7) | 26.1 (5.5)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.99, t-test, 2 sided

10. Secondary Outcome: Mean Total Bilirubin Value
Description: Mean Total Bilirubin value between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
mg/dL | 7.1 (1.0) | 1.1 (1.7)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.39, t-test, 2 sided

11. Secondary Outcome: Mean Lactate Dehydrogenase Value
Description: Mean Lactate Dehydrogenase (LDH) value between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: unit/L
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
unit/L | 323.9 (254.1) | 253.7 (323.9)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.43, t-test, 2 sided

12. Secondary Outcome: Mean Adult Hemoglobin Percentage
Description: Mean Adult Hemoglobin (HbA) percentage between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: % of Adult Hemoglobin (HbA)
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
% of Adult Hemoglobin (HbA) | 2.8 (6.9) | 59.6 (8.2)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p < 0.01, t-test, 2 sided

13. Secondary Outcome: Mean Sickle Hemoglobin Percentage
Description: Mean Sickle Hemoglobin (HbS) Percentage between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: % of Sickle Hemoglobin (HbS)
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
% of Sickle Hemoglobin (HbS) | 68.7 (17.1) | 36.7 (7.5)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.01, t-test, 1 sided

14. Secondary Outcome: Mean Fetal Hemoglobin Percentage
Description: Mean Fetal Hemoglobin (HbF) Percentage between Sickle Cell Disease Pre-transplantation and Sickle Cell Disease Post-Transplantation
Time Frame: as for outcome 1
Population: Pre-specified in the protocol to only assess this Outcome Measure in the Sickle Cell Disease Arms/Groups.
Measure: Mean (Standard Deviation); unit: % of Fetal Hemoglobin
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation
Number analyzed (Participants) | 6 | 5
% of Fetal Hemoglobin | 10.4 (9.1) | .5 (.8)
Statistical Analysis 1: Comparison: Sickle Cell Disease Pre-Transplantation vs Sickle Cell Disease Post-Transplantation; Test type: Other; p = 0.04, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 6 months
Description: All Grade 2 and above adverse events (AE) that are related to diagnostic and interventions directly related to this study whether volunteered by the participant, discovered by study personnel during questioning, or detected through physical examination, clinically significant laboratory test, or other means will be recorded.
Arm/Group | Sickle Cell Disease Pre-Transplantation | Sickle Cell Disease Post-Transplantation | Sickle Cell Trait (HbAS) | HbAA (Healthy Volunteers)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/3
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/7 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/77/NCT04476277/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT04476277/ICF_001.pdf